CLINICAL TRIAL: NCT03987295
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AL001 in Heterozygous Carriers of Granulin or C9orf72 Mutations Causative of Frontotemporal Dementia
Brief Title: A Phase 2 Study to Evaluate Safety of Long-term AL001 Dosing in Frontotemporal Dementia (FTD) Patients (INFRONT-2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alector Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL001-2
Record Dates: First submitted 2019-05-14; First posted 2019-06-17 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Granulin and C9orf72 (Experimental): IV administration of AL001; 60 mg/kg, every 4 weeks [q4w]
  Interventions: Drug: AL001

INTERVENTIONS:
Drug: AL001 — 60 mg/kg of AL001 every 4 weeks

SUMMARY:
A Phase 2 open label study evaluating the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of AL001 in participants with a Granulin mutation or C9orf72 mutation causative of frontotemporal dementia.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open label study evaluating the safety, tolerability, PK and PD of AL001 administered intravenously in participants with a Granulin mutation or C9orf72 mutation causative of frontotemporal dementia.

ELIGIBILITY:
Inclusion Criteria:

* At screening, female participants must be nonpregnant and nonlactating
* In good physical health on the basis of no clinically significant findings from medical history, physical examinations (PEs), laboratory tests, ECGs, and vital signs.
* Participant is a carrier of a loss of function progranulin gene (GRN) mutation or carrier of a hexanucleotide repeat expansion C9orf72 mutation

Exclusion Criteria:

* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* History of alcohol abuse or substance abuse
* Participant resides in a skilled nursing facility, convalescent home, or long term care facility

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ljubenkov, MD, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (4):
  - UCSF, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Glenn Biggs Institute for Alzheimer's and Neurodegenerative Diseases UT Health San Antonio, San Antonio, Texas
- Canada (2):
  - Lawson Health Research Institute, St. Joseph's, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Germany (2):
  - Technical University of Munich, München
  - University of Ulm, Ulm
- University of Brescia, Brescia, Italy
- Netherlands (2):
  - Brain Research Center - PPDS, Amsterdam
  - Erasmus University Medical Center, Rotterdam
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- aFTD-GRN: aFTD-GRN - asymptomatic frontotemporal dementia with heterozygous progranulin gene mutation
  Part 1 - Latozinemab administered intravenously (60 mg/kg, every 4 weeks [q4w]), for a total of 25 doses (96-week dosing period); Part 2 - Latozinemab administered intravenously (60 mg/kg, every 4 weeks [q4w]), for a total of 25 doses (96-week dosing period).
- FTD-GRN: FTD-GRN - symptomatic carriers of GRN mutation causative of FTD
  Part 1 - Latozinemab administered intravenously (60 mg/kg, every 4 weeks [q4w]), for a total of 25 doses (96-week dosing period); Part 2 - Latozinemab administered intravenously (60 mg/kg, every 4 weeks [q4w]), for a total of 25 doses (96-week dosing period).
- FTD-C9orf72: FTD-C9orf72 - symptomatic carriers of C9orf72 hexanucleotide repeat expansion mutation causative of FTD
  Part 1 - Latozinemab administered intravenously (60 mg/kg, every 4 weeks [q4w]), for a total of 25 doses (96-week dosing period); Part 2 - Latozinemab administered intravenously (60 mg/kg, every 4 weeks [q4w]), for a total of 25 doses (96-week dosing period).
Period: Overall Study
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Started | 5 | 12 | 16
Completed | 5 | 5 | 6
Not Completed | 0 | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72 | Total
Number analyzed (Participants) | 5 | 12 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 11 | 23
  >=65 years | 0 | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 59.0 [32 to 63] | 59.5 [48 to 78] | 60.0 [40 to 74] | 59.0 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 9 | 14
  Male | 4 | 8 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 10 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 10 | 16 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Severity of TEAEs
Description: Number of TEAEs categorized by severity
Time Frame: 197 weeks
Population: There is no statistical analysis for this primary end point.
Measure: Number; unit: TEAEs (all)
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 12 | 16
TEAEs (all)
  Mild | 43 | 58 | 84
  Moderate | 4 | 9 | 24
  Severe | 3 | 1 | 4
  Life Threatening | 0 | 0 | 0
  Death | 0 | 0 | 1

2. Primary Outcome: Severity of Treatment-Related TEAEs
Description: Number of treatment-related TEAEs categorized by severity
Time Frame: 197 weeks
Population: There is no statistical analysis for this primary end point.
Measure: Number; unit: TEAEs (treatment-related)
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 12 | 16
TEAEs (treatment-related)
  Mild | 5 | 1 | 12
  Moderate | 1 | 1 | 5
  Severe | 0 | 0 | 0
  Life Threatening | 0 | 0 | 0
  Death | 0 | 0 | 0

3. Primary Outcome: Any TEAE Leading to Study Drug Discontinuation
Description: Number of TEAEs leading to study drug discontinuation
Time Frame: 197 weeks
Population: There is no statistical analysis for this primary end point.
Measure: Number; unit: TEAE leading to discontinuation
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 12 | 16
TEAE leading to discontinuation | 0 | 1 | 1

4. Primary Outcome: Immunogenicity Antidrug Antibodies (ADA) Titer
Description: Titer values of antidrug antibodies (ADAs) in participants receiving latozinemab at week 97/Part 1 end of study
Time Frame: 97 weeks
Population: There is no statistical analysis for this primary end point.
Measure: Median (Full Range); unit: Titers
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 12 | 16
Titers
  Week 2 - ADA Titer | 320.0 [20 to 5120] | 20.0 [20 to 2560] | 40.0 (0.00) [20 to 160]
  Week 13 - ADA Titer | 160.0 [20 to 2560] | 160.0 [160 to 640] | 120.0 [80 to 160]
  Week 25 - ADA Titer | 320.0 [320 to 320] | 330.0 [20 to 640] | 80.0 [20 to 160]
  Week 37 - ADA Titer | 0 [0 to 0] | 80.0 [20 to 320] | 90.0 [20 to 160]
  Week 49 - ADA Titer | 0 [0 to 0] | 320.0 [40 to 640] | 20.0 [20 to 20]
  Week 61 - ADA Titer | 0 [0 to 0] | 0 [0 to 0] | 160.0 [160 to 160]
  Week 73 - ADA Titer | 0 [0 to 0] | 160.0 [160 to 160] | 0 [0 to 0]
  Week 85 - ADA Titer | 0 [0 to 0] | 160.0 [160 to 160] | 20.0 [20 to 20]
  Week 97 - ADA Titer | 20.0 [20 to 20] | 0 [0 to 0] | 160.0 [160 to 160]

5. Primary Outcome: Confirmatory Immunogenicity Antidrug Antibodies (ADA) Responses
Description: Presence of confirmatory antidrug antibodies (ADAs) in participants who test positive for ADA at week 97 (Part 1 End of Study).
Time Frame: 97 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 5 | 9
Participants
  ADA Positive | 1 | 0 | 2
  ADA Negative | 4 | 5 | 7

6. Primary Outcome: Change From Baseline in Sheehan Suicidality Tracking Scale
Description: The Sheehan Suicidality Tracking Scale (S-STS) is a structured assessment tool used to evaluate the presence, severity, and frequency of suicidal ideation and behavior. It includes items that address passive thoughts of death, active suicidal ideation, intent, planning, suicide attempts, and non-suicidal self-injury. The S-STS total score ranges from 0 to 64, based on 16 items each rated from 0 (not at all) to 4 (extremely), with higher scores indicating greater severity of suicidal ideation, intent, or behavior. The total score provides a quantitative measure of suicidality severity and is sensitive to change over time, making it suitable for clinical monitoring and research use.
Time Frame: 197 weeks
Population: There is no statistical analysis for this primary endpoint.
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 1 | 3
Scores | 0 (0) | 0 | 0 (0)

7. Secondary Outcome: Longitudinal Percent Change From Baseline of CSF PGRN
Description: The percent change from baseline to specified timepoints of PGRN in CSF. The baseline visit is labeled as week 1 and therefore the 96th week is labeled as week 97.
Time Frame: 97 weeks
Population: There is no statistical analysis for this secondary end point.
Measure: Mean (Standard Deviation); unit: percent change of ug/L
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 4 | 8 | 11
percent change of ug/L
  Week 49 | 198.16 (110.255) | 104.05 (103.349) | 101.61 (38.492)
  Week 97: number analyzed (Participants) | 4 | 2 | 6
  Week 97 | 189.46 (113.802) | 59.73 (24.034) | 144.73 (54.994)

8. Secondary Outcome: Longitudinal Percent Change From Baseline in Plasma PGRN
Description: The percent change from baseline to specified timepoints for PGRN in plasma. The baseline visit is labeled as week 1 and therefore the 96th week is labeled as week 97.
Time Frame: 97 weeks
Population: There is no statistical analysis for this secondary end point.
Measure: Mean (Standard Deviation); unit: percent change in ug/L
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 12 | 16
percent change in ug/L
  Week 49: number analyzed (Participants) | 5 | 8 | 11
  Week 49 | 177.39 (51.352) | 151.32 (59.321) | 178.82 (58.406)
  Week 97: number analyzed (Participants) | 5 | 5 | 9
  Week 97 | 185.37 (43.763) | 188.12 (47.847) | 157.93 (92.695)

9. Secondary Outcome: Longitudinal Levels of Sortilin in WBCs
Description: The overall change from baseline in Sortilin in WBCs.
Time Frame: 97 weeks
Population: WBC samples for analysis for Sortilin expression were collected to serve as a pharmacodynamic biomarker of target engagement. Development of this assay found that stability of these samples was not reliable for accurate measurement. Hence, we did not measure Sortilin in this study.
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Latozinemab Concentration in Serum
Description: Serum concentration of Latozinemab at week 97.
Time Frame: 97 weeks
Population: There is no statistical analysis for this secondary end point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 2 | 7
ng/mL | 236000 (69100) | 250000 (24700) | 265000 (77000)

11. Secondary Outcome: Cmax of Latozinemab at Specified Timepoints
Description: Maximum observed concentration of Latozinemab at week 96 of treatment.
Time Frame: 97 weeks
Population: There is no statistical analysis for this secondary end point.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 2 | 7
ug/mL | 1810 (352) | 1320 (255) | 1510 (145)

12. Secondary Outcome: Ctrough of Latozinemab at Specified Timepoints
Description: Trough concentration of Latozinemab at week 96 of treatment
Time Frame: 97 weeks
Population: There is no statistical analysis for this secondary endpoint.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 2 | 14
ug/mL | 236 (69.1) | 250 (24.7) | 252 (66.7)

13. Secondary Outcome: ARCmax of Latozinemab
Description: Ratio of latozinemab Cmax at week 61 to the Cmax at week 1
Time Frame: 61 weeks
Population: There is no statistical analysis for this endpoint.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
Number analyzed (Participants) | 5 | 8 | 10
Ratio | 1.22 (0.192) | 1.23 (0.236) | 1.39 (0.712)

ADVERSE EVENTS:
Time Frame: 197 weeks
Arm/Group | aFTD-GRN | FTD-GRN | FTD-C9orf72
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12 | 1/16
Serious Adverse Events (participants affected / at risk) | 1/5 | 3/12 | 2/16
Other Adverse Events (participants affected / at risk) | 4/5 | 9/12 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aFTD-GRN (N=5) | FTD-GRN (N=12) | FTD-C9orf72 (N=16)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aFTD-GRN (N=5) | FTD-GRN (N=12) | FTD-C9orf72 (N=16)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Crying (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site paraesthesia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Illusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Impulsive behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Device physical property issue (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 7 (7)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parkinsonian rest tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 5 (5)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 6 (6)
Viral rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study had the following limitations:

* No placebo control arm
* Small number of participants
* A high number of participants discontinued the study due to disease progression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alector's agreements with principal investigators may vary but will not prohibit any investigator from publishing. Alector supports the publication of the results from all centers in a multi-center trial, and its agreements include provisions to enable the multi-center publication to occur before publication of data from a single site.

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03987295/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT03987295/SAP_001.pdf